CLINICAL TRIAL: NCT06060899
Title: Intraoperative Blood Loss Under Standard Versus Low Pneumoperitoneum Pressure During Laparoscopic Liver Resection: Study Protocol for a Randomized Controlled Trial
Brief Title: Intraoperative Blood Loss Under Standard Versus Low Pneumoperitoneum Pressure During Laparoscopic Liver Resection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Jagiellonian University (Other); Regional Oncology Center, Białystok, Poland (Unknown)
Responsible Party: Principal Investigator, Wacław Hołówko, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB/160/2022
Record Dates: First submitted 2023-08-26; First posted 2023-09-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Liver Tumor
Keywords: laparoscopic liver resection; pneumoperitoneum pressure; blood loss
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard pneumoperitoneum pressure (Active Comparator): Laparoscopic liver resection performed in standard (14mmHg) pneumoperitoneum pressure
  Interventions: Procedure: Pneumoperitoneum 14mmHg
- Low pneumoperitoneum pressure (Experimental): Laparoscopic liver resection performed in low (10mmHg) pneumoperitoneum pressure
  Interventions: Procedure: Pneumoperitoneum 10mmHg

INTERVENTIONS:
Procedure: Pneumoperitoneum 14mmHg — Performing surgery in 14mmHg pneumoperitoneum pressure
  Arms: Standard pneumoperitoneum pressure
Procedure: Pneumoperitoneum 10mmHg — Performing surgery in 10mmHg pneumoperitoneum pressure
  Arms: Low pneumoperitoneum pressure

SUMMARY:
Commonly the pressure of about 14 mmHg is applied during laparoscopic liver resection (LLR) with moderate neuromuscular blockade. Lowering the pneumoperitoneum pressure combined with deep neuromuscular blockade may sustain optimal operating space with providing better short-term postoperative results. It has been proved in randomized controlled trials in colorectal or bariatric patients, however there is lack of similar data for laparoscopic liver resection. Doubts about lowering the pneumoperitoneum pressure too hasty are supported by apprehension of worse bleeding control during liver parenchyma transection and its impact on postoperative results.

The aim of the trial is to assess the impact of standard (14 mmHg; arm 1) versus low (10 mmHg; arm 2) pneumoperitoneum pressure on intraoperative blood loss, what will be the primary outcome. As secondary endpoints following outcomes will be measured: quality of operating space, intraoperative adverse events, quality of recovery, postoperative renal function, 30-day postoperative complications rate, length of hospital stay. The investigators assume that lower pneumoperitoneum provides non-inferior blood loss control during laparoscopic liver resection with better postoperative results.

DETAILED DESCRIPTION:
After signing the informed consent patients will be randomized into 2 groups. Randomization will be conducted by investigators via drawing a sealed envelope with computer-generated intervention code at the Department just before patient transfer to the operating theatre. There will be two study arms with 1:1 fashion

For both trial arms additional routine elements of perioperative anesthesia care will be defined:

* low central vein pressure, aimed for 5 ± 2 mmHg with restrictive fluid therapy
* ventilation in a volume-controlled mode without intraoperative high positive end-expiratory pressure (PEEP)
* invasive arterial blood pressure monitoring with maintaining mean arterial pressure ≥ 60 mmHg
* maintaining hemoglobin concentration > 8g/dl
* maintaining normothermia and normoglycemia
* maintaining oxygenation >94%, in case of hypercapnia with respiratory acidosis, the respiratory rate and tidal volume will be stepwise increased

The surgeon will be blinded to the study arm and level of pneumoperitoneum pressure.

The blood loss during liver parenchyma transection and total procedure blood loss will be reported based on the amount of sucked outside intraperitoneal fluids after liver transection and after procedure without volume inserted for intraperitoneal irrigation. The estimated blood loss will be measured in milliliters. Patients who are converted to open surgery are excluded from the analysis of the primary end-point.

During the procedure, the surgeon will be asked regularly to rate the quality of operating space in accordance to the Leiden Surgical Rating Scale. In case of inadequate operating space, pneumoperitoneum pressure may be increased by 2 mmHg (with maximum of 16 mmHg in arm 1. and 12 mmHg in arm 2.). Intraoperative adverse events will be assessed in accordance to ClassIntra classification. Quality of recovery (QoR) will be measured on postoperative day 1, 3 and 5 with patient reported QoR-40 questionnaire, 30-day postoperative complication rate will be assessed in accordance to Clavien-Dindo classification. Length of hospital stay will be counted from the date of surgery to the discharge day. All patients will be followed up by researchers who are blinded to the intraoperative grouping.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to perform elective laparoscopic major liver resection
* Age of 18 years or older
* Signed informed consent

Exclusion Criteria:

* Severe cardiopulmonary disease
* Severe renal disease
* Liver cirrhosis
* Emergency surgery
* Pregnancy
* Patient's refusal of participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | Intraoperative
  Intraoperative blood loss in ml

SECONDARY OUTCOMES:
Quality of the operating space | Intraoperative
  Expressed in accordance to Leiden scale (L-SRS) and the rate of need for increase of pneumoperitoneum pressure
  Score 1-5 (where 1 means extremely poor conditions; 5- optimal conditions)
  From multiple measurements, value submitted for analysis will be the lowest reported during the surgery.
Intraoperative adverse events | Intraoperative
  Expressed in accordance to ClassIntra scale
  Grades 0-V (where 0 means no deviation; V- intraoperative death of the patient)
Quality of postoperative rehabilitation | Postoperative day 1, Postoperative day 3, Postoperative day 5
  Expressed in accordance to questionaire QoR-40
  40 questions with 1-5 points each (total score minimum 40 points; maximum 200 points)
Risk of postoperative complications | 30 postoperative days
  Expressed in accordance to Clavien-Dindo classification in 30-day postoperative period
Length of hospital stay | From date of surgery until the date of disscharge or date of death from any cause, whichever came first, assessed up to 100 days
  Expressed in days

CONTACTS AND LOCATIONS:
Overall Officials: Wacław Hołówko, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of General, Transplant and Liver Surgery, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Protocol will be published in a journal
Supporting Information: Study Protocol
Time Frame: 31/12/2023
Access Criteria: Open access